CLINICAL TRIAL: NCT04999215
Title: Choline-PET: Exploratory Study Assessing the Potential Role of F-choline PET Imaging in New and Emerging Indications
Acronym: F-choline
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-9489
Record Dates: First submitted 2021-08-05; First posted 2021-08-10 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Lesion With Known or Suspected F-choline Uptake
Keywords: Imaging; F-choline PET; Diagnostic performance
MeSH Terms: interventions — fluorocholine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main arm (Experimental): F-choline intravenous injection
  Interventions: Drug: F-choline intravenous injection

INTERVENTIONS:
Drug: F-choline intravenous injection — Participants will receive one injection of F-choline before undergoing hybrid PET/CT imaging per standard procedures. F-choline PET examinations may be repeated, if this judged to be in the patient's best interest by his referring physician and the study staff, up to a maximum 4 examinations per year.
  Other Names: Fluorocholine

SUMMARY:
Choline is an important building block of phospholipids in cell membranes. Certain cancers and medical conditions are known to demonstrate increased absorption and incorporation of choline into their cell membranes. 18-F-fluorocholine (F-choline) and 11-C-choline (C-choline) are diagnostic positron emission tomography (PET) radiotracers that can be used to image, in vivo, the metabolism of choline. Both tracers have been extensively studied in prostate cancer and C-choline has obtained US FDA approval for the investigation of recurrent prostate cancer. F-choline is currently not approved for clinical use by the FDA or Health Canada, but it offers many advantages over C-choline due to its better physical characteristics (mainly due to its positron range, shorter and longer half-life). In recent years, reports have started to emerge on broader potential applications of choline PET imaging, particularly for imaging parathyroid adenomas, certain cervical cancers and certain liver cancers.

The main objective is to discover and explore potential new and emerging indications in which F-choline could play a role and provide clinically relevant information.

Secondary objectives are 1) To assess the safety of F-choline PET imaging using F-choline produced at the CRCHUM; 2) assess changes in patient/disease management following F-choline PET imaging.

Researchers hypothesize that F-choline will provide useful and incremental clinical information in a variety of conditions, and outperform the "standard" workup in numerous conditions.

F-Choline PET exams will be performed on hybrid PET/CT scanners according to standard procedures. These examinations could be repeated at the discretion of the treating physician (up to a maximum of 4 exams per year) if the treating physician and the research team deem this could provide additional clinically useful information (for example, by helping to assess response to newly started therapy).

The results will be provided to the attending physician and any new knowledge could lead to a change in treatment or an investigation of the condition that prompted enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a known or suspected condition in which F-choline PET imaging might provide clinically useful information.

Exclusion Criteria:

* Pregnancy
* Breastfeeding woman, unwilling to discontinue breastfeeding for 48 hours
* Known allergy to F-choline or any excipients
* Pediatric patient (< 18 years old)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2032-07-01 (Estimated); Study Completion 2032-08-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance (sensitivity and specificity) of F-choline PET/CT | 3 months
  "Gold-standard" will be a composite of other imaging modalities, pathological data when available, and clinical follow-up.
Adverse reaction to the F-choline injection | 24 hours
  Absence or presence of adverse reactions related to F-choline injection (yes or no)

SECONDARY OUTCOMES:
Change in management following F-choline PET/CT | 3 months
  Frequency of change in management, comparing planned management before and after F-choline PET/CT

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Juneau, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'université de Montréal, Montreal, Quebec, Canada